CLINICAL TRIAL: NCT00098865
Title: A Phase II Pilot Study Of Thalidomide With Temozolomide In Patients With Relapsed Or Progressive Brain Tumors Or Neuroblastoma
Brief Title: Thalidomide and Temozolomide in Relapsed or Progressive CNS Disease or Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Boston Children's Hospital (Other); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Mark W. Kieran, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-279 DFCI; P30CA006516 (NIH); CDR0000396780 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-09

CONDITIONS: Central Nervous System Tumor, Pediatric; Neuroblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma | interventions — Temozolomide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide and Temozolomide (Experimental): Thalidomide:
  Oral thalidomide on days 1-28 of a 28 day cycle initiated at 3 mg/kg and increased to maximum dose of 24 mg/kg or 1000 mg as tolerated.
  Temozolomide:
  Oral temozolomide on days 1-5 of 28 day cycle given at 200 mg/m2 or 150 mg/m2 for patients who had previously received significant therapy to the bone marrow (chemotherapy or radiation) or cranial spinal radiation.
  Patients were treated for 6 cycles unless disease progression or excessive toxicity. Treatment could continue beyond 6 cycles if absent disease progression
  Interventions: Drug: temozolomide; Drug: thalidomide

INTERVENTIONS:
Drug: temozolomide — The lower 150/m2 Temozolomide dose was for patients who had previously received significant therapy to the bone marrow (chemotherapy or radiation) or cranial spinal raditation.
  Other Names: Temodar
Drug: thalidomide — Calculated dose was rounded down to the nearest 50mg, or up to 50mg if calculated dose was less than 50mg. Patients increased the daily dose by 50mg (one capsule) on a weekly basis unitl either unacceptable toxicity or a maximum dose.
  Other Names: Thalamid

SUMMARY:
RATIONALE: Thalidomide may stop the growth of tumor cells by stopping blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining thalidomide with temozolomide may kill more tumor cells.

PURPOSE: This phase II trial is studying the effectiveness of combining thalidomide with temozolomide in treating young patients who have relapsed or progressive brain tumors or recurrent neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of thalidomide and temozolomide in pediatric patients with relapsed or progressive poor prognosis brain tumors or recurrent neuroblastomas.

Secondary

* Determine preliminarily evidence of biologic activity of this regimen in these patients.
* Determine the toxic effects of this regimen in these patients.

STATISTICAL DESIGN: The primary data analysis will estimate the percentage of patients who can complete 6 months of therapy in the mixed population. With a target accrual of 20 patients the 90% confidence for the true feasibility rate will be no wider than 40%.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* diagnosis of 1 of the following:

  * Poor prognosis brain tumor

    * Relapsed or progressive disease
    * No curative therapy exists
  * Neuroblastoma

    * Recurrent disease NOTE: *Histologic confirmation not required for brain stem glioma; patients with brain stem glioma must have clinical and radiographic evidence of disease
* Patients with brain stem glioma must have symptoms lasting < 3 months comprising cranial nerve deficits (often VI or VII) and/or ataxia and/or long tract signs

PATIENT CHARACTERISTICS:

Age

* 21 and under

Performance status

* Karnofsky 50-100% OR
* Lansky 50-100%

Life expectancy

* More than 2 months

Hematopoietic

* Hemoglobin ≥ 9.0 g/dL
* Platelet count > 75,000/mm^3
* WBC > 2,000/mm^3
* Absolute neutrophil count > 1,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* SGOT and SGPT ≤ 2 times normal (SGOT ≤ 4 times normal for patients taking Zantac)
* Alkaline phosphatase ≤ 2 times normal
* No active hepatic disease ≥ grade 3

Renal

* Creatinine < 1.5 mg/dL OR
* Creatinine clearance ≥ 70 mL/min
* No active renal disease ≥ grade 3

Cardiovascular

* No active cardiac disease ≥ grade 3

Pulmonary

* No active pulmonary disease ≥ grade 3

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation

  * Willing and able to participate in the System for Thalidomide Education and Prescription Safety (S.T.E.P.S.^®) program
* No active psychiatric disease ≥ grade 3

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed

  * No prior thalidomide

Chemotherapy

* Prior chemotherapy allowed

  * No prior temozolomide

Endocrine therapy

* Concurrent steroids allowed

Radiotherapy

* Prior radiotherapy allowed

Surgery

* Prior surgery allowed

Other

* Concurrent antiseizure medications allowed
* No other concurrent investigational agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2002-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Kieran, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 patients were enrolled between 2002 to 2007 at the Dana-Farber Cancer Institute.
Pre-assignment Details: For pediatric patients with relapsed or progressive brain tumors and neuroblastoma.
Period: Overall Study
Arm/Group | Thalidomide and Temozolomide
Started | 15
Completed | 6
Not Completed | 9
Not completed — Progressive Disease | 6
Not completed — Adverse Event | 2
Not completed — Alternative Therapy | 1

BASELINE CHARACTERISTICS:
Population: The analysis population represents all enrolled and treated patients.
Arm/Group | Thalidomide and Temozolomide
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 15
Disease Type [Number; unit: participants]
  Brain Tumor | 8
  Neuroblastoma | 7

OUTCOME MEASURES:

1. Primary Outcome: Therapy Completion Rate
Description: Feasibility in this study was defined as completion of 6 months of thalidomide with temozolomide therapy. The corresponding therapy completion rate is defined as the proportion of patients who completed 6 months of therapy.
Time Frame: 6 months
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Thalidomide and Temozolomide: Thalidomide:
  Oral thalidomide on days 1-28 of a 28 day cycle initiated at 3 mg/kg and increased to maximum dose of 24 mg/kg or 1000 mg as tolerated.
  Temozolomide:
  Oral temozolomide on days 1-5 of 28 day cycle given at 200 mg/m2 or 150 mg/m2 for patients who had previously received significant therapy to the bone marrow (chemotherapy or radiation) or cranial spinal radiation.
  Patients were treated for 6 cycles unless disease progression or excessive toxicity. Treatment could continue beyond 6 cycles if absent disease progression
  temozolomide: The lower 150/m2 Temozolomide dose was for patients who had previously received significant therapy to the bone marrow (chemotherapy or radiation) or cranial spinal raditation.
  thalidomide: Calculated dose was rounded down to the nearest 50mg, or up to 50mg if calculated dose was less than 50mg. Patients increased the daily dose by 50mg (one capsule) on a weekly basis unitl either unacceptable toxicity or a maximum dose.
Arm/Group | Thalidomide and Temozolomide
Number analyzed (Participants) | 15
proportion of participants | .40 [.19 to .64]

2. Secondary Outcome: Overall Response
Description: Overall response is the best response during 6 months of therapy measured by radiographic response.
  Complete Response (CR): Disappearance of all detectable tumors by imaging, if initially positive, as well as 2 consecutively negative CSF cytologic examinations (if the initial cytology was positive).
  Partial Response (PR): > 50% reduction in the sum of the products of the maximum perpendicular diameter of all measurable lesions; or 2 consecutively negative CSF cytologies and a < 50% reduction in tumor size.
  Stable Disease (SD): < 50% reduction in the sum of the products of the maximum perpendicular diameters of all measurable lesions, and persistently negative or positive CSF cytology Progressive Disease (PD): > 25% increase in the size of any measurable lesion, the appearance of a new radiographically demonstrable lesion, or the conversion of negative CSF cytology to positive, as confirmed by at least one repeat CSF cytology
Time Frame: Assessed every 8 weeks while on treatment and every 3 months for one year off-study
Measure: Number; unit: participants
Arm/Group | Thalidomide and Temozolomide
Number analyzed (Participants) | 15
participants
  Partial Response | 1
  Stable Disease | 9
  Progressive Disease | 4
  Unevaluable | 1

3. Secondary Outcome: Overall Survival
Description: Time from registration to death. Patients alive at last follow-up were censored.
Time Frame: Assessed after treatment discontinued every 3 months up to 2 years.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide and Temozolomide
Number analyzed (Participants) | 15
months | 12.8 [6.7 to 41.2]

ADVERSE EVENTS:
Time Frame: Clinical assessment of drug toxicities was performed every clinic visit including CBC and serum biochemistries were collected every 2 weeks for the first 8 weeks of therapy and then monthly.
Groups:
- Thalidomide and Temzolomide: Thalidomide:
  Oral thalidomide on days 1-28 of a 28 day cycle initiated at 3 mg/kg and increased to maximum dose of 24 mg/kg or 1000 mg as tolerated.
  Temozolomide:
  Oral temozolomide on days 1-5 of 28 day cycle given at 200 mg/m2 or 150 mg/m2 for patients who had previously received significant therapy to the bone marrow (chemotherapy or radiation) or cranial spinal radiation.
  Patients were treated for 6 cycles unless disease progression or excessive toxicity. Treatment could continue beyond 6 cycles if absent disease progression.
Arm/Group | Thalidomide and Temzolomide
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide and Temzolomide (N=15)
Hemoglobin (Blood and lymphatic system disorders) | 2
Hematologic-other (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Vision-blurred (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Infection w/ unk ANC catheter related (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Leukocytes (Investigations) | 4
Lymphopenia (Investigations) | 2
Neutrophils (Investigations) | 5
Platelets (Investigations) | 4
ALT, SGPT (Investigations) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide and Temzolomide (N=15)
Hemoglobin (Blood and lymphatic system disorders) | 8
Cardiac-other (Cardiac disorders) | 2
Hearing-other (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Abdomen, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Fever w/o neutropenia (General disorders) | 3
Rigors/chills (General disorders) | 1
Constitutional, other (General disorders) | 3
Pain-other (General disorders) | 1
Infection-other (Infections and infestations) | 1
Leukocytes (Investigations) | 9
Lymphopenia (Investigations) | 5
Neutrophils (Investigations) | 6
Platelets (Investigations) | 7
Alkaline phosphatase (Investigations) | 2
ALT, SGPT (Investigations) | 8
AST, SGOT (Investigations) | 6
Creatinine (Investigations) | 3
Bicarbonate (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Neuropathy-motor (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 1
Euphoria (Psychiatric disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less